CLINICAL TRIAL: NCT04089358
Title: StepByStep: A Randomized Trial of a Mobile Health and Social Media Physical Activity Intervention Among Adolescent and Young Adult Childhood Cancer Survivors
Brief Title: Mobile Health and Social Media Physical Activity Intervention Among Adolescent and Young Adult Childhood Cancer Survivors, the StepByStep Study
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: MedStar Georgetown University Hospital (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ALTE2031; NCI-2020-01916 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ALTE2031 (Other: Children's Oncology Group); COG-ALTE2031 (Other: DCP); ALTE2031 (Other: CTEP); U01CA246665 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2019-09-10; First posted 2019-09-13 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Organizational Objectives; Health Promotion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (educational materials, Fitbit) (Active Comparator): Participants receive educational materials about physical activity and wear a Fitbit daily for 48 weeks.
  Interventions: Other: Educational Intervention; Device: FitBit
- Intervention group (educational materials, goal set, Fitbit) (Experimental): See outline
  Interventions: Other: Educational Intervention; Device: FitBit; Other: Goal Setting; Other: Health Promotion and Education; Other: Media Intervention; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Educational Intervention — Receive educational materials
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Device: FitBit — Wear a Fitbit
Other: Goal Setting — Set goals
  Arms: Intervention group (educational materials, goal set, Fitbit)
Other: Health Promotion and Education — Receive text message about goal setting
  Arms: Intervention group (educational materials, goal set, Fitbit)
Other: Media Intervention — Follow Instagram group
  Arms: Intervention group (educational materials, goal set, Fitbit)
Behavioral: Telephone-Based Intervention — Receive phone call about goal setting
  Arms: Intervention group (educational materials, goal set, Fitbit)

SUMMARY:
This phase III trial compares a multi-component mobile health and social media physical activity intervention versus wearing a physical activity tracker alone among adolescent and young adult childhood cancer survivors. Regular physical activity helps maintain healthy weight, energy levels, and health. Adolescents and young adults who complete treatment for cancer are often less active. They may gain weight and have more health problems compared to people the same age who have not had treatment for cancer. Comparing the 2 programs will help researchers learn how to increase physical activity levels over time and also how changes in physical activity levels affect health and quality of life over time.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effects of a multi-component physical activity intervention including a Fitbit, individualized goal setting, and a social media peer support group compared to the control condition (Fitbit only) on physical activity among adolescent and young adult survivors of childhood cancer (AYA survivors) who do not meet physical activity guidelines.

SECONDARY OBJECTIVES:

I. To evaluate the effects of a multi-component physical activity intervention including a Fitbit, individualized goal setting, and a social media peer support group compared to the control condition (Fitbit only) on biomarkers predictive of cardiometabolic health among adolescent and young adult survivors of childhood cancer (AYA survivors) who do not meet physical activity guidelines.

II. To evaluate the effects of a multi-component physical activity intervention including a Fitbit, individualized goal setting, and a social media peer support group compared to the control condition (Fitbit only) on health-related quality of life among adolescent and young adult survivors of childhood cancer (AYA survivors) who do not meet physical activity guidelines.

OUTLINE: Participants are randomized to 1 of 2 groups.

INTERVENTION GROUP: Participants receive educational materials about physical activity.

INTENSIVE PHASE (24 WEEKS): Participants wear a physical activity tracker (Fitbit) daily as well as receiving weekly reminders from study staff to wear it. They also receive goal setting sessions each week (by text, phone call, etc.) to set personalized step count goals using the Fitbit application (app). Lastly, participants receive an invitation to follow and post on an online social media peer support group (Instagram), where study staff provide encouraging advice and messages about physical activity 2-3 times per week, announce badges/awards every week, and moderate a forum to discuss physical activity and use of the Fitbit.

MAINTENANCE PHASE (24 WEEKS): Participants wear a Fitbit daily but do not receive reminders to wear it. They also set their own step count goals weekly and check in with study staff monthly for assistance with goal setting. Participants take the lead posting content on the Instagram account moderated by the study staff. Study staff only post once per week with general physical activity-related questions and provide no badges.

CONTROL GROUP: Participants receive educational materials about physical activity and wear a Fitbit daily for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* First diagnosis of malignant neoplasm (International Classification of Diseases for Oncology [ICD-O] behavior code of "3") in first and continuous remission at the time of enrollment
* Curative cancer treatment must have included chemotherapy (including cellular therapy) and/or radiation (including radioactive iodine)

  * Note: Childrens Oncology Group (COG) therapeutic trial participation is not required
* All cancer treatment must have been completed within 3-36 calendar months prior to enrollment
* Patients must have a life expectancy of > 1 year
* Self-report of < 420 minutes of moderate-to-vigorous physical activity per week as assessed via the study-specific Physical Activity Worksheet

  * Note: See COG Study Web Page for the Godin-Shephard Leisure Time Physical Activity Questionnaire or link to online calculator
* Ambulatory and no known medical contraindications to increasing physical activity

  * Note: Patients with amputation, rotationplasty, or other prothesis are not automatically excluded as long as they are ambulatory and have no known medical contraindications to increasing physical activity and all other eligibility criteria are satisfied
* No known significant physical or cognitive impairment that would prevent use of the electronic devices used for the protocol intervention (e.g. Fitbit, smartphone, tablet, or computer)
* Able to read and write English

  * Note: For patients < 18 years, consenting parent/legal guardian does not have to be able to read and write English
* All patients and/or their parents or legal guardians must sign a written informed consent

  * Note: Informed consent may be obtained electronically/online if allowed by local site policy and Institutional Review Board (IRB)/Research Ethics Board (REB) of record
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Post-menarchal female patients who are pregnant or planning to become pregnant in the next year are excluded

  * Note: Pregnancy status can be established by clinical history with patient. Post-menarchal female patients are eligible as long as they agree to use an effective contraceptive method (including abstinence) during study participation
* Patients with previous hematopoietic stem cell transplant (HSCT) are excluded

  * Note: Patients with previous autologous HSCT, chimeric antigen receptor T-cell (CAR T-cell) therapy, and other cellular cancer therapies can participate as long as all other eligibility criteria are satisfied

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 387 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in minutes of moderate-to-vigorous physical activity (MVPA) per day from Baseline Evaluation | 12 months
  Moderate-to-vigorous physical activity (MVPA) will be tracked using a wearable activity monitor (research-grade accelerometer) that counts how often (how many times) someone performs MVPA over a 7 day period. Total minutes above the moderate-intensity threshold will be divided by the number of valid days to obtain minutes of MVPA per day.

SECONDARY OUTCOMES:
Cardiopulmonary fitness | 12 months
  Cardiopulmonary fitness is an objective biomarker of exercise capacity and will be assessed by the 2-Minute Step Test. During the 2-Minute Step Test, participants are asked to march in place as quickly as possible for 2 minutes. This test requires a stopwatch and a counter. Stopping, starting, and resting during the test are allowed as needed. Steps are counted.
Body mass index (BMI) | 12 months
  Self-reported height and weight will be collected from the participants prior to the participant initiating the 2-Minuite Step Test. BMI will be calculated as weight (kg) divided by height squared (m2). BMI will be examined as a potential covariate for the analysis of fitness as measured by the 2-Minute Step Test.
Resting heart rate | 12 months
  Resting heart rate will be taken using the Fitbit physical activity tracker heart rate monitor prior to the participant initiating the 2-Minute Step Test.
Health-related quality of life (HRQOL) | 12 months
  HRQOL will be measured with the Pediatric Quality of Life inventory (PedsQL) 4.0 Generic Core Scales (global functioning, physical functioning, and social functioning scales, specifically) and the 18-item PedsQL 4.0 Multidimensional Fatigue Scale, which encompasses three subscales: (1) general fatigue (6 items), (2) sleep/rest fatigue (6 items), and (3) cognitive fatigue (6 items).115-118 Questions refer to how much of a problem each item was during the past month. Items are reverse-scored and transformed to a scale from 0-100, in which higher scores indicate better HRQOL.
Total cholesterol | 12 months
  A dried blood sample will be collected on each participant after a minimum of an 8-hour fast. A total of 3 drops of blood will be collected by finger stick with a lancet. Samples will be tested for: total cholesterol.
High density lipoprotein (HDL) | 12 months
  A dried blood sample will be collected on each participant after a minimum of an 8-hour fast. A total of 3 drops of blood will be collected by finger stick with a lancet. Samples will be tested for: high density lipoprotein (HDL).
Low density lipoprotein (LDL) | 12 months
  A dried blood sample will be collected on each participant after a minimum of an 8-hour fast. A total of 3 drops of blood will be collected by finger stick with a lancet. Samples will be tested for: low density lipoprotein (LDL).
Triglycerides | 12 months
  A dried blood sample will be collected on each participant after a minimum of an 8-hour fast. A total of 3 drops of blood will be collected by finger stick with a lancet. Samples will be tested for: triglycerides.
Glucose | 12 months
  A dried blood sample will be collected on each participant after a minimum of an 8-hour fast. A total of 3 drops of blood will be collected by finger stick with a lancet. Samples will be tested for: glucose.
Insulin (HOMA-IR) | 12 months
  A dried blood sample will be collected on each participant after a minimum of an 8-hour fast. A total of 3 drops of blood will be collected by finger stick with a lancet. Samples will be tested for: insulin.
Hemoglobin A1c (HbA1c) | 12 months
  A dried blood sample will be collected on each participant after a minimum of an 8-hour fast. A total of 3 drops of blood will be collected by finger stick with a lancet. Samples will be tested for: hemoglobin A1c (HbA1c).
High sensitivity C-reactive protein (CRP) | 12 months
  A dried blood sample will be collected on each participant after a minimum of an 8-hour fast. A total of 3 drops of blood will be collected by finger stick with a lancet. Samples will be tested for: high sensitivity C-reactive protein (CRP).

CONTACTS AND LOCATIONS:
Overall Officials: Nina S Kadan-Lottick, Principal Investigator — Children's Oncology Group
Locations (116):
- United States (114):
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Palms West Radiation Therapy, Loxahatchee Groves, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Vannie Cook Children's Clinic, McAllen, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - IWK Health Centre, Halifax, Nova Scotia

REFERENCES:
- [Derived] Beight LJ, Mendoza JA, Leisenring WM, Collier W, Olsen ME, Ross WL, Santiago-Rivera Y, Bryant S, Rotatori J, Ness KK, Hurtado-de-Mendoza A, Baker KS, Chow EJ, Kadan-Lottick NS. Design and methods of the StepByStep randomized trial of a mobile health and social media physical activity intervention among adolescent and young adult survivors of childhood cancer: A report from the Children's Oncology Group. Contemp Clin Trials. 2024 Oct;145:107645. doi: 10.1016/j.cct.2024.107645. Epub 2024 Jul 28. PMID 39079612